CLINICAL TRIAL: NCT05879796
Title: A Controlled Clinical Study of Envafolimab (PD-L1 Antibody) Subcutaneous Injection Combined With Endostar and Concurrent Chemoradiotherapy in Treatment of Locally Advanced Primary Cervical Cancer
Brief Title: Envafolimab Combined With Endostar and Concurrent Chemoradiotherapy for Locally Advanced Primary Cervical Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2023108
Record Dates: First submitted 2023-05-19; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Radiation; Brachytherapy; envafolimab; Endostatins; endostar protein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- envafolimab combined with endostar and concurrent chemoradiotherapy: Concurrent Chemoradiation； Envafulimab,150mg, subcutaneous, QW. Maintenance therapy until disease progression, or intolerable toxicity, or up to 1 year; Endostar, administered at a dose of 75 mg/day, QW, was administered by intravenous pump on day 1 of each cycle, and the first dose was administered on the first day of radiotherapy, 6 cycles in total.
  Interventions: Drug: cis-platinum; Radiation: radiation; Drug: Envafolimab Injection; Drug: Recombinant Human Endostatin Injection
- concurrent chemoradiotherapy: Concurrent Chemoradiation:
  Cisplatin 40 mg/m2, day1, 7 days as a cycle, 6 cycles in total; External beam radiotherapy was performed using IMRT/VMAT radiotherapy with pelvic and/or extended field irradiation at a total dose of 45-50.4 Gy;1.8-2.0 Gy/f,25- 28 f. In patients with pelvic lymph node metastasis, para-aortic lymph node metastasis, and retroperitoneal lymph node metastasis, local lesions were simultaneously boosted to 60 Gy. In FIGO stage IIIB, simultaneous or late course boost to 60 Gy was given parametrially.
  Brachytherapy: High dose rate (HDR) afterloading brachytherapy was used, with a total dose of 30-40 Gy and a cumulative dose of 80-85 Gy at point A/HRCTV D90; if the tumor diameter was ≥ 4cm, the cumulative dose of ≥ 87 Gy at point A/HRCTV D90. Brachytherapy combined with external beam radiation therapy was completed within 8 weeks.
  Interventions: Drug: cis-platinum; Radiation: radiation

INTERVENTIONS:
Drug: cis-platinum — chemotherapeutics
  Other Names: Cisplatin
Radiation: radiation — External beam radiotherapy was performed using IMRT/VMAT radiotherapy with pelvic and/or extended field irradiation at a total dose of 45-50.4 Gy;1.8-2.0 Gy/f,25 -28 f. In patients with pelvic lymph node metastasis, para-aortic lymph node metastasis, and retroperitoneal lymph node metastasis, local lesions were simultaneously boosted to 60 Gy. In FIGO stage IIIB, simultaneous or late course boost to 60 Gy was given parametrially.
  Brachytherapy: High dose rate (HDR) afterloading brachytherapy was used, with a total dose of 30-40 Gy and a cumulative dose of 80-85 Gy at point A/HRCTV D90; if the tumor diameter was ≥ 4 cm, the cumulative dose of ≥ 87 Gy at point A/HRCTV D90. Brachytherapy combined with external beam radiation therapy was completed within 8 weeks.
  Other Names: External beam radiotherapy; Brachytherapy
Drug: Envafolimab Injection — PD-L1 antibody
  Other Names: KN035
  Groups: envafolimab combined with endostar and concurrent chemoradiotherapy
Drug: Recombinant Human Endostatin Injection — angiogenesis inhibitors
  Other Names: endostar
  Groups: envafolimab combined with endostar and concurrent chemoradiotherapy

SUMMARY:
The goal of this study is to determine efficacy and safety of envafolimab combined with Endostar and concurrent chemoradiation in the treatment of locally advanced primary cervical cancer.

Thirty participants will be divided into control group (n = 15) and experimental group (n = 15). The control group received concurrent chemoradiation, and the experimental group received envafolimab combined with endostar and concurrent chemoradiation.

DETAILED DESCRIPTION:
This study was a single-center, prospective cohort study. Thirty Participants will be non-randomized in a 1:1 ratio divided into control group (n = 15) and experimental group (n = 15).

The control group: chemoradiation;

The experimental group: envafolimab combined with endostar and concurrent chemoradiation.

Concurrent chemoradiation:

Cisplatin 40 mg/m2, day1, 7 days as a cycle, 6 cycles in total; External beam radiotherapy was performed using IMRT/VMAT radiotherapy with pelvic and/or extended field irradiation at a total dose of 45-50.4 Gy;1.8-2.0 Gy/f,25- 28 f. In patients with pelvic lymph node metastasis, para-aortic lymph node metastasis, and retroperitoneal lymph node metastasis, local lesions were simultaneously boosted to 60 Gy. In FIGO stage IIIB, simultaneous or late course boost to 60 Gy was given parametrially.

Brachytherapy: High dose rate (HDR) afterloading brachytherapy was used, with a total dose of 30-40 Gy and a cumulative dose of 80-85 Gy at point A/HRCTV D90; if the tumor diameter was ≥ 4cm, the cumulative dose of ≥ 87 Gy at point A/HRCTV D90. Brachytherapy combined with external beam radiation therapy was completed within 8 weeks.

Envafulimab,150mg, subcutaneous, QW. Maintenance therapy until disease progression, or intolerable toxicity, or up to 1 year; Endostar, administered at a dose of 75 mg/day, QW, was administered by intravenous pump on day 1 of each cycle, and the first dose was administered on the first day of radiotherapy, 6 cycles in total.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed advanced cervical cancer， FIGO 2018 clinical stages IB3/IIA2 with positive para-aortic lymph nodes 、IIB-IVA disease, patients with locally advanced cervical cancer who are judged by their physician to be eligible for concurrent chemoradiotherapy in this trial, and have not received treatment before enrollment;
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Expected life > 3 months
* LVEF≥55%
* Adequate bone marrow, hepatic and renal function including the following:

Haemoglobin ≥ 90g/L, absolute neutrophil count ≥ 1,500 /µL, platelets ≥100,000 /µL; Serum creatinine ≤ 1.5 x ULN; Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2.5 x ULN or ≤ 5 x ULN in the presence of liver metastases;total bilirubin ≤ 1.5 x ULN or patients with Gilbert 's syndrome who can have total bilirubin≤ 2.5 x ULN

* Patients of childbearing potential must agree to use effective contraception during the trial, and have a negative serum or urine pregnancy test
* Non-lactating patients
* Signed informed consent

Exclusion Criteria:

* Prior treatment with an anti-PD-1, anti-PD-L1 or anti-vascular agents
* Any previous abdominal or pelvic radiotherapy
* Patients with other invasive malignancies within the last 5 years
* Serious uncontrolled medical conditions that, in the opinion of the investigator, would compromise the subject 's ability to receive treatment with the study protocol, such as concurrent serious medical conditions, including serious heart disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension, uncontrolled infection, active peptic ulcer, etc.
* Receipt of other experimental agents or participation in another clinical study for anticancer therapeutic purposes within 30 days of first dose
* Serious infection occurred within 4 weeks before the start of study treatment, including but not limited to infectious complications requiring hospitalization, bacteremia or severe pneumonia
* Patients who are known to be human immunodeficiency virus (HIV) positive
* Patients who are hepatitis B surface antigen positive (HBsAg), and whose peripheral blood hepatitis B virus deoxyribonucleic acid (HBV-DNA) titer is ≥ 1 ×103IU/mL; if HBsAg is positive, and peripheral blood HBV-DNA is < 1 ×103 IU/mL, the subject is eligible if the investigator believes that the subject has stable chronic hepatitis B and will not increase the risk of the subject;
* Hepatitis C virus (HCV) antibody positive or human immunodeficiency virus (HIV) antibody positive, and HCV RNA test positive
* Patients judged unsuitable for this study by the investigator

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be selected with the help of oncologists in Peking university third hospital. All participants are advanced cervical cancer.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-05-16 (Estimated); Primary Completion 2024-05-16 (Estimated); Study Completion 2026-05-16 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | From Baseline to 2 years
  ORR was assessed by the site Investigator using RECIST 1.1 and was defined as the percentage of patients with a confirmed overall response of CR or PR.

SECONDARY OUTCOMES:
Disease control rate | From Baseline to 2 years
  DCR was assessed by the site Investigator using RECIST 1.1 and was defined as the percentage of patients with a confirmed overall response of CR or PR or SD.
progression-free survival | From Baseline to 2 years
  the time of all participants from the start of the treatment to tumor progression
overall survival | From Baseline to 2 years
  the time from the start of the treatment to the death of any cause.
The adverse events according to NCI-CTCAE v5.0 | From the start of treatment until 30 days after the last study drug administration
  Safety (according to NCI-CTCAE v5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Ping Jiang, MD, Principal Investigator — Study Principal Investigator

IPD SHARING:
Plan to Share IPD: No